CLINICAL TRIAL: NCT04407234
Title: The Impact of Tirzepatide on Gastric Emptying (GE) in Overweight/Obese Non-diabetic Subjects and in Overweight/Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Measure Stomach Emptying in Overweight Non-diabetic and Diabetic Participants Using Tirzepatide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17376; I8F-MC-GPHU (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-04

CONDITIONS: Overweight; Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — Tirzepatide; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tirzepatide + Acetaminophen (Experimental): Participants received 5mg tirzepatide on Day 1 and Day 8; 10 mg tirzepatide on Day 15, 22 and 29; 15 mg tirzepatide on Day 36 administered subcutaneously (SC) and 160 mg acetaminophen administered orally on Day -1, Day 2 and Day 37.
  Interventions: Drug: Tirzepatide; Drug: Acetaminophen

INTERVENTIONS:
Drug: Tirzepatide — Tirzepatide administered SC.
  Other Names: LY3298176
Drug: Acetaminophen — Acetaminophen administered orally.

SUMMARY:
The purpose of this study is to learn more about how tirzepatide affects stomach emptying in overweight/very overweight participants. Participants include those without diabetes and those with type 2 diabetes.

The study will last about 13 weeks for each participant, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 27 to 45 kilograms per meter squared (kg/m²), inclusive at screening
* For nondiabetic subjects: as determined by medical history, physical examination, and safety assessments at screening
* For participants with a confirmed type 2 diabetes diagnosis: The condition must be managed either by diet and exercise alone or on a stable dose of metformin for the past 3 months
* Willing and agreeable to commit to the duration of the study and undergo study procedures as instructed by the clinic staff

Key Exclusion Criteria

* Have undergone gastric bypass or bariatric surgery
* Have received prescription drugs or over the counter drugs that promote weight loss in the past 6 months prior to screening
* For participants with a confirmed type 2 diabetes diagnosis: Have experienced more than 1 episode of severe low blood sugar that require emergency treatment, hospitalization or third parties to administer rescue treatment, in the past 6 months
* Have any lifetime history of a suicide attempt
* Have other medical conditions or medical history that make participation in the study unsafe or which may interfere in the interpretation of the results of the study
* Unwilling to comply with smoking and alcohol restrictions during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Clinical Pharmacology of Miami, Hialeah, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://trials.lillytrialguide.com/en-US/trial/2VTN9N9xaJ4FhSAZuwJdif?conditionId=1wecF0AgauDdWnqHV7GJGP

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Diabetic: Participants received 5 milligrams (mg) tirzepatide on Day 1 and Day 8; 10 mg tirzepatide on Day 15, 22 and 29; 15 mg tirzepatide on Day 36 administered subcutaneously (SC) and 160 mg acetaminophen administered orally on Day -1, Day 2 and Day 37.
- Type 2 Diabetes Mellitus (T2DM): Participants received 5mg tirzepatide on Day 1 and Day 8; 10 mg tirzepatide on Day 15, 22 and 29; 15 mg tirzepatide on Day 36 administered SC and 160 mg acetaminophen administered orally on Day -1, Day 2 and Day 37.
Period: Overall Study
Arm/Group | Non-Diabetic | Type 2 Diabetes Mellitus (T2DM)
Started | 18 | 18
Received at Least One Dose of Study Drug | 18 | 18
Completed | 15 | 15
Not Completed | 3 | 3
Not completed — Adverse Event | 3 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Non-Diabetic; T2DM: Participants received 5 mg tirzepatide on Day 1 and Day 8; 10 mg tirzepatide on Day 15, 22 and 29; 15 mg tirzepatide on Day 36 administered SC and 160 mg acetaminophen administered orally on Day -1, Day 2 and Day 37.
- Total: Total of all reporting groups
Arm/Group | Non-Diabetic | T2DM | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (10.8) | 56.2 (5.5) | 50.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 18 | 36
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 14 | 16 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration [ AUC(0-tlast)] of Acetaminophen
Description: Area Under the Concentration Time Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration [ AUC(0-tlast)] of Acetaminophen
Time Frame: Pre-dose, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12, 24 and 36 hours post-dose on Day 1, Day 2 and Day 37 , Day 2 and Day 37
Population: All randomized participants who received at least one dose of acetaminophen and have evaluable acetaminophen PK data.
Measure: Geometric Mean (90% Confidence Interval); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- Reference:160 mg Acetaminophen (Day -1): Participants received 160 mg acetaminophen administered orally on Day -1.
- Test: 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2): Participants received 5 mg tirzepatide on Day 1 and Day 8 and 160 mg acetaminophen administered orally Day 2.
- Test: 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37): Participants received 15 mg tirzepatide on Day 36 administered SC and 160 mg acetaminophen administered orally on Day 37.
Arm/Group | Reference:160 mg Acetaminophen (Day -1) | Test: 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2) | Test: 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37)
Number analyzed (Participants) | 36 | 36 | 30
nanograms*hours per milliliter (ng*h/mL) | 49384 [43635 to 55890] | 43523 [38456 to 49257] | 57049 [50171 to 64869]
Statistical Analysis 1: Comparison: Reference:160 mg Acetaminophen (Day -1) vs Test: 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2); Test type: Superiority; Wilcoxon signed rank test; Ratio of geometric least squares mean = 0.881, 90% CI 2-sided [0.803 to 0.967]
Statistical Analysis 2: Comparison: Reference:160 mg Acetaminophen (Day -1) vs Test: 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37); Test type: Superiority; Wilcoxon signed rank test; Ratio of geometric least squares mean = 1.16, 90% CI 2-sided [1.05 to 1.28]

2. Primary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of Acetaminophen
Description: Maximum Observed Drug Concentration (cmax) of Acetaminophen
Time Frame: Pre-dose, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12, 24 and 36 hours post-dose on Day 1, Day 2 and Day 37 , Day 2 and Day 37
Population: All randomized participants who received at least one dose of acetaminophen and have evaluable acetaminophen PK data.
Measure: Geometric Mean (90% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Groups:
- Test: 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37: Participants received 15 mg tirzepatide on Day 36 administered SC and 160 mg acetaminophen administered orally on Day 37.
Arm/Group | Reference:160 mg Acetaminophen (Day -1) | Test: 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2) | Test: 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37
Number analyzed (Participants) | 36 | 36 | 30
nanograms per milliliter (ng/mL) | 11925 [10566 to 13460] | 5314 [4708 to 5998] | 8099 [7111 to 9225]
Statistical Analysis 1: Comparison: Reference:160 mg Acetaminophen (Day -1) vs Test: 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2); Test type: Superiority; Wilcoxon signed rank test; Ratio of geometric least squares mean = 0.446, 90% CI 2-sided [0.390 to 0.509]
Statistical Analysis 2: Comparison: Reference:160 mg Acetaminophen (Day -1) vs Test: 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37; Test type: Superiority; Wilcoxon signed rank test; Ratio of geometric least squares mean = 0.679, 90% CI 2-sided [0.589 to 0.783]

3. Secondary Outcome: Hemoglobin A1c (HbA1c) Data by Diabetic Status
Description: Levels of Hemoglobin A1c (HbA1c) were assessed at predose on Day 29, and at follow-up (Day 64).
Time Frame: Predose on Day 29 and follow-up (Day 64)
Population: All participants who received at least one dose of acetaminophen or tirzepatide, whether or not they completed all protocol requirements
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Groups:
- Non-Diabetic; T2DM: Participants received 5mg tirzepatide on Day 1 and Day 8; 10 mg tirzepatide on Day 15, 22 and 29; 15 mg tirzepatide on Day 36 administered SC and 160 mg acetaminophen administered orally on Day -1, Day 2 and Day 37.
Arm/Group | Non-Diabetic | T2DM
Number analyzed (Participants) | 15 | 15
Percentage of HbA1c
  Day 29 ± 1 | 5.37 (0.45) | 7.27 (0.79)
  Day 64 ± 1 (Follow-Up) | 5.29 (0.45) | 6.87 (0.75)

4. Secondary Outcome: PK: Area Under the Concentration Time Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration [ AUC(0-tlast)] of Acetaminophen at Steady State For Non-diabetic
Description: Area Under the Concentration Time Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration [ AUC(0-tlast)] of Acetaminophen at Steady State For Non-diabetic
Time Frame: Pre-dose, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12, 24 and 36 hours post-dose on Day 1, Day 2 and Day 37 , Day 2 and Day 37
Population: All participants who received at least one dose of acetaminophen and have evaluable acetaminophen PK data.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- Reference (Non-diabetic):160 mg Acetaminophen (Day -1): Participants received 160 mg acetaminophen administered orally on Day -1.
- Test (Non-diabetic): 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2): Participants received 5 mg tirzepatide on Day 1 and Day 8 and 160 mg acetaminophen administered orally Day 2.
- Test (Non-diabetic): 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37): Participants received 15 mg tirzepatide on Day 36 administered SC and 160 mg acetaminophen administered orally on Day 37
Arm/Group | Reference (Non-diabetic):160 mg Acetaminophen (Day -1) | Test (Non-diabetic): 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2) | Test (Non-diabetic): 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37)
Number analyzed (Participants) | 18 | 18 | 15
nanograms*hours per milliliter (ng*h/mL) | 44350 [37276 to 52766] | 39389 [33107 to 46864] | 54735 [45695 to 65563]
Statistical Analysis 1: Comparison: Reference (Non-diabetic):160 mg Acetaminophen (Day -1) vs Test (Non-diabetic): 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2); Test type: Superiority; Ratio of geometricleast squares mean = 0.888, 90% CI 2-sided [0.778 to 1.01]
Statistical Analysis 2: Comparison: Reference (Non-diabetic):160 mg Acetaminophen (Day -1) vs Test (Non-diabetic): 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37); Test type: Superiority; Ratio of geometricleast squares mean = 1.23, 90% CI 2-sided [1.07 to 1.42]

5. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration [ AUC(0-tlast)] of Acetaminophen at Steady State For T2DM
Description: Area Under the Concentration Versus Time Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration [ AUC(0-tlast)] of Acetaminophen at Steady State For T2DM
Time Frame: Pre-dose, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12, 24 and 36 hours post-dose on Day 1, Day 2 and Day 37 , Day 2 and Day 37
Population: All participants who received at least one dose of acetaminophen and have evaluable acetaminophen PK data.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- Reference (T2DM):160 mg Acetaminophen (Day -1): Participants received 160 mg acetaminophen administered orally on Day -1.
- Test (T2DM): 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2): Participants received 5 mg tirzepatide on Day 1 and Day 8 and 160 mg acetaminophen administered orally Day 2.
- Test (T2DM): 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37): Participants received 15 mg tirzepatide on Day 36 administered SC and 160 mg acetaminophen administered orally on Day 37
Arm/Group | Reference (T2DM):160 mg Acetaminophen (Day -1) | Test (T2DM): 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2) | Test (T2DM): 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37)
Number analyzed (Participants) | 18 | 18 | 15
nanograms*hours per milliliter (ng*h/mL) | 54989 [46219 to 65424] | 48090 [40420 to 57215] | 59440 [49623 to 71199]
Statistical Analysis 1: Comparison: Reference (T2DM):160 mg Acetaminophen (Day -1) vs Test (T2DM): 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2); Test type: Superiority; Ratio of geometricleast squares mean = 0.875, 90% CI 2-sided [0.766 to 0.999]
Statistical Analysis 2: Comparison: Reference (T2DM):160 mg Acetaminophen (Day -1) vs Test (T2DM): 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37); Test type: Superiority; Ratio of geometricleast squares mean = 1.08, 90% CI 2-sided [0.938 to 1.25]

6. Secondary Outcome: PK: Cmax of Acetaminophen at Steady State Non-diabetic
Description: PK: Cmax of Acetaminophen at Steady State Non-diabetic
Time Frame: Pre-dose, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12, 24 and 36 hours post-dose on Day 1, Day 2 and Day 37 , Day 2 and Day 37
Population: All participants who received at least one dose of acetaminophen and have evaluable acetaminophen PK data.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Arm/Group | Reference (Non-diabetic):160 mg Acetaminophen (Day -1) | Test (Non-diabetic): 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2) | Test (Non-diabetic): 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37)
Number analyzed (Participants) | 18 | 18 | 15
nanograms per milliliter (ng/mL) | 10255 [8680 to 12115] | 4646 [3932 to 5489] | 8245 [6891 to 9866]
Statistical Analysis 1: Comparison: Reference (Non-diabetic):160 mg Acetaminophen (Day -1) vs Test (Non-diabetic): 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2); Test type: Superiority; Ratio of geometricleast squares mean = 0.453, 90% CI 2-sided [0.376 to 0.545]
Statistical Analysis 2: Comparison: Reference (Non-diabetic):160 mg Acetaminophen (Day -1) vs Test (Non-diabetic): 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37); Test type: Superiority; Ratio of geometricleast squares mean = 0.804, 90% CI 2-sided [0.660 to 0.979]

7. Secondary Outcome: PK: Cmax of Acetaminophen at Steady State For T2DM
Description: PK: Cmax of Acetaminophen at Steady State T2DM
Time Frame: Pre-dose, 0.5, 0.75, 1, 2, 3, 4, 6, 9, 12, 24 and 36 hours post-dose on Day 1, Day 2 and Day 37 , Day 2 and Day 37
Population: All participants who received at least one dose of acetaminophen and have evaluable acetaminophen PK data.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Arm/Group | Reference (T2DM):160 mg Acetaminophen (Day -1) | Test (T2DM): 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2) | Test (T2DM): 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37)
Number analyzed (Participants) | 18 | 18 | 15
nanograms per milliliter (ng/mL) | 13868 [11738 to 16385] | 6078 [5144 to 7181] | 7954 [6648 to 9517]
Statistical Analysis 1: Comparison: Reference (T2DM):160 mg Acetaminophen (Day -1) vs Test (T2DM): 5 mg Tirzepatide + 160 mg Acetaminophen (Day 2); Test type: Superiority; Ratio of geometricleast squares mean = 0.438, 90% CI 2-sided [0.364 to 0.527]
Statistical Analysis 2: Comparison: Reference (T2DM):160 mg Acetaminophen (Day -1) vs Test (T2DM): 15 mg Tirzepatide + 160 mg Acetaminophen (Day 37); Test type: Superiority; Ratio of geometricleast squares mean = 0.574, 90% CI 2-sided [0.471 to 0.698]

ADVERSE EVENTS:
Time Frame: Baseline Up To 45 Days
Description: All participants who received at least one dose of study drug.
Arm/Group | Non-diabetic | T2DM
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 16/18 | 16/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-diabetic (N=18) | T2DM (N=18)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 6 (6) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 14 (19)
Vomiting (Gastrointestinal disorders) | 3 (4) | 7 (16)
Chills (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 16 (16) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT04407234/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT04407234/SAP_001.pdf